CLINICAL TRIAL: NCT01100554
Title: Upper Airway Collapsibility Evaluation in Different Sedative Levels by Sleep Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Yung-Lun Ni, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 980717A3
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Bronchoscopy; Obstructive Sleep Apnea; Conscious Sedation
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Consciousness Monitors; Electroencephalography; Electromyography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- all patients (Experimental)
  Interventions: Device: Sleep endoscopy

INTERVENTIONS:
Device: Sleep endoscopy — Conscious sedation will be done under intravenous propofol infusion. The sedative level would be monitored and adjusted accord to the Bispectral Index monitor. After the adequate sedative level is achieved, a bronchoscopy (Olympus, BF) was inserted from the right nostril. The velopharynx, oropharynx, larynx, and hypopharynx obstructions were evaluated.
  Other Names: Bispectral Index; electroencephalograms(EEG); electromyograms(EMG)

SUMMARY:
The purpose of this study is to evaluate the upper airway collapsibility by sleep endoscopy in different sedative levels. Propofol pump infusion will be used to achieve conscious sedation. Bispectral Index monitor will be applied to the monitor the conscious level. Two different sedative levels (BIS 65-75, 50-60) will be achieved for upper airway evaluation. The severities of upper airway obstruction will be evaluated the correlation to the disease severities. Mandible advancement will be done to evaluate the response for oral appliance.

DETAILED DESCRIPTION:
Obstructive sleep apnea/hypopnea syndrome (OSAHS) is a disorder characterized by recurrent upper airway collapse during sleep. Clinical consequences as increased cardiovascular events and automobile accidents were noted. Polysomnography is diagnostic while continuous positive airway pressure (CPAP) is the standard treatment. The adherence of CPAP treatment remained suboptimal, between 29 to 83%. In selected cases, alternative treatments were considered useful. However, how to choose candidates is still an issue.

Sleep endoscopy has been introduced since 1991 to allow direct visualization of the upper airway under sleep simulation. It predicts better outcome in non-adherent OSAHS patients who received alternative treatment. However, the ideal dose, drug, and sedative depth were not known.

Bispectral Index (BIS) monitor is a noninvasive neurophysiological monitoring device that been introduced since late 1990's. By applying a sensor to the forehead, the BIS obtained electroencephalograms(EEG) and electromyograms(EMG) which were transformed into simplified scaled numbers through 0-100. It has been applied in the real time monitor of anesthesia depth during operation or recovery, monitor of sleep in critical illness patients and gastrointestinal endoscopy sedation.

This study focuses on CPAP non-adherent patients. It evaluates the upper airway collapsibility in awake and two different sedative levels, BIS 65-75 (light sedation) and BIS 50-60(deep sedation). Conscious sedation will be achieved by propofol pump infusion. No benzodiazepam or opioid are used to avoid the effect of upper airway muscle tone and respiratory drive. The patency over the velopharynx, oropharynx, larynx, and hypopharynx will be recorded. Specific obstruction patterns such as tongue base retraction, epiglottis anterior-posterior decent, omega-shaped epiglottis,and bilateral arytenoids anterior drawing will also be recorded. The correlation of the upper airway collapsibility between sedative depth and sleep stages (ex. NREM vs. REM) will be evaluated. Besides, mandible advancement will be done under deep sedation. The response will guide further treatment choice for those CPAP non-adherent patient.

ELIGIBILITY:
Inclusion Criteria:

* Normal volunteer: cases with no sleep apnea symptoms and AHI<5
* Study cases: CPAP non-adherent sleep apnea patient

Exclusion Criteria:

* ASA > 3
* allergy to propofol, xylocaine, or food (egg, bean, milk)
* congestive heart failure
* severe obstructive airway disease
* head injury, seizure, cerebrovascular accident history
* age < 18 year-old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Upper airway collapsibility
  The severity of upper aiwray collapses in different sedative levels will be evaluated by the sleep endoscopy. The correlation between the disease severities and airway collapsibilities will be evaluated.

SECONDARY OUTCOMES:
Mandible advancement response and oral appliance response | 6 month and 1 year after oral appliance
  Patients with response to mandible advancement will be referred to oral appliance to treat OSA. The treatment outcome will be followed.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Lun Lo, MD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Department or Thoracic Medicine, Chang Gung Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Kotecha BT, Hannan SA, Khalil HM, Georgalas C, Bailey P. Sleep nasendoscopy: a 10-year retrospective audit study. Eur Arch Otorhinolaryngol. 2007 Nov;264(11):1361-7. doi: 10.1007/s00405-007-0366-1. Epub 2007 Jun 20. PMID 17579877
- [Background] Bachar G, Feinmesser R, Shpitzer T, Yaniv E, Nageris B, Eidelman L. Laryngeal and hypopharyngeal obstruction in sleep disordered breathing patients, evaluated by sleep endoscopy. Eur Arch Otorhinolaryngol. 2008 Nov;265(11):1397-402. doi: 10.1007/s00405-008-0637-5. Epub 2008 Mar 8. PMID 18327599
- [Derived] Lo YL, Ni YL, Wang TY, Lin TY, Li HY, White DP, Lin JR, Kuo HP. Bispectral Index in Evaluating Effects of Sedation Depth on Drug-Induced Sleep Endoscopy. J Clin Sleep Med. 2015 Sep 15;11(9):1011-20. doi: 10.5664/jcsm.5016. PMID 25979098